CLINICAL TRIAL: NCT01929993
Title: Large Loop Excision of Transformation Zone Cone Versus Straight Wire Excision of Transformation Zone : Histopathological Analysis of Excision Margins
Brief Title: A Trial of Two Electrosurgical Conizations: Histopathological Analysis of Excision Margins
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oswaldo Cruz Foundation (Other)
Responsible Party: Principal Investigator, MJCamargo, PHD, Oswaldo Cruz Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 522/12
Record Dates: First submitted 2012-06-10; First posted 2013-08-28 (Estimated); Results first posted 2015-06-09 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-06

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Conization; Cervical Intraepithelial Neoplasia; Cervix Dysplasia; Therapy; Electrosurgery
MeSH Terms: conditions — Uterine Cervical Dysplasia; Hyperthermia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SWETZ (Experimental): Straight wire excision of transformation zone is an electrosurgical conization method, which uses a straight wire electrode.
  Interventions: Procedure: SWETZ
- LLETZ cone (Active Comparator): LLETZ cone is a electrosurgical conization method, which is performed with a large loop electrode of 20 mm depth.
  Interventions: Procedure: LLETZ cone

INTERVENTIONS:
Procedure: SWETZ — Straight wire excision of transformation zone is an electrosurgical conization method, which uses a straight wire electrode as a knife to remove the dysplastic epithelium of the cervix.
  Other Names: NETZ - Needle excision of transformation zone
  Arms: SWETZ
Procedure: LLETZ cone — LLETZ cone is a electrosurgical conization method, which is performed with a large loop electrode of 20 mm depth. The loop is applied to the cervix outside the lateral margin of the transformation zone and brought slowly to the controlateral transformation zone margin.
  Other Names: LEEP - Loop electrosurgical excision procedure.
  Arms: LLETZ cone

SUMMARY:
The purpose of this trial is to evaluate if Straight Wire Excision of the Transformation Zone (SWETZ) is superior to (Large Loop Excision of the Transformation Zone) LLETZ cone in reducing the incomplete excision of disease.

DETAILED DESCRIPTION:
Cone biopsy is a surgical procedure which objectives the excision of endocervical pre-invasive disease located at transformation zone or glandular epithelium. Although cone biopsy is considered adequate for the treatment of endocervical dysplastic epithelium , using electrosurgery as opposed to the cold knife technique of cone biopsy has been criticized because of the perceived potential for incomplete excision of disease, thermal damage and surgical specimen fragmentation, which might increase the risk of missing early invasive cancer. Also, incomplete excision margin of disease exposes women to an increased risk of residual post-treatment disease.

The standard procedure, Large Loop Excision of the Transformation Zone (LLETZ-cone), is performed with a large loop electrode of 20-25 mm depth.

The experimental intervention is Straight Wire Excision of the Transformation Zone (SWETZ), a method of excision using a 1cm straight disposal of 0.20 wire to remove the endocervical transformation zone or glandular disease.

Both procedures were previously studied in another clinical trial(NCT00995020), but the histological analysis were inconclusive for many outcomes. SWETZ were superior to LLETZ cone to acquire complete excision of disease, with no statistical significance, probably due to the small sample size.

This study objectives a better histological analyses of the surgical specimens related to incomplete excision, thermal damage and fragmentation.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible if the colposcopist decided that a cone biopsy was indicated.
* Common indications for a cone biopsy included:

  * High-grade Squamous Intraepithelial Lesion in a type 3 transformation zone,
  * suspicion of micro-invasive or invasive carcinoma and
  * suspicion of glandular disease.

Exclusion Criteria:

* Patients were excluded if pregnancy, coagulation disorders and cervicitis were present or if they refused to participate in the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria J Camargo, PHD, Study Director — Oswaldo Cruz Foundation
Locations (1):
- Fernandes Figueira Institute - Oswaldo Cruz Foundation, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Russomano F, Tristao MA, Cortes R, de Camargo MJ. A comparison between type 3 excision of the transformation zone by straight wire excision of the transformation zone (SWETZ) and large loop excision of the transformation zone (LLETZ): a randomized study. BMC Womens Health. 2015;15:12. doi: 10.1186/s12905-015-0174-5. Epub 2015 Feb 18. PMID 25783647

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women who needed type 3 excision of the Transformation Zone referred to a colposcopy clinic in Rio de Janeiro, Brazil, after cytological screening between January 2008 thru December 2011.
Groups:
- Straight Wire Excision of Transformation Zone (SWETZ): Straight wire excision of transformation zone is an electrosurgical conization method, which uses a straight wire electrode to remove the dysplastic epithelium of the cervix.
- Large Loop Excision of the Transformation Zone (LLETZ-cone): Large Loop Excision of the Transformation Zone (LLETZ-cone) is a electrosurgical conization method, which is performed with a large loop electrode of 20 mm depth. The loop is applied to the cervix outside the lateral margin of the transformation zone and brought slowly to the controlateral transformation zone margin.
Period: Overall Study
Arm/Group | Straight Wire Excision of Transformation Zone (SWETZ) | Large Loop Excision of the Transformation Zone (LLETZ-cone)
Started | 82 | 82
Completed | 52 | 54
Not Completed | 30 | 28
Not completed — Protocol Violation | 4 | 6
Not completed — Absent CIN, invasion present or artifact | 26 | 22

BASELINE CHARACTERISTICS:
Groups:
- Straight Wire Excision of Transformation Zone (SWETZ): Straight wire excision of transformation zone (SWETZ) is an electrosurgical conization method, which uses a straight wire electrode as a knife to remove the dysplastic epithelium of the cervix.
- Total: Total of all reporting groups
Arm/Group | Straight Wire Excision of Transformation Zone (SWETZ) | Large Loop Excision of the Transformation Zone (LLETZ-cone) | Total
Number analyzed (Participants) | 52 | 54 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (13.3) | 42.3 (10.7) | 43.1 (12.0)
Sex/Gender, Customized [Number; unit: participants]
  Female | 52 | 54 | 106

OUTCOME MEASURES:

1. Primary Outcome: The Prevalence of Incomplete Excision of Dysplasia at the Endocervical Excision Margin as Recognized Histologically.
Description: Incomplete excision was considered when high-grade intraepithelial (CIN2-3) or microinvasive neoplasia was present in the endocervical limit of the excised specimen.
Time Frame: one month after the procedure
Population: Any compromised margin.
Measure: Number; unit: participants
Arm/Group | SWETZ | LLETZ Cone
Number analyzed (Participants) | 52 | 54
participants | 28 | 39

ADVERSE EVENTS:
Time Frame: Adverse events were observed during or through the first week after the procedures.
Description: Participants at risk: the ones originally included and who received one of the procedures, no matter who had been excluded from the primary outcome analysis.
Arm/Group | SWETZ | LLETZ Cone
Serious Adverse Events (participants affected / at risk) | 1/81 | 1/78
Other Adverse Events (participants affected / at risk) | 1/81 | 1/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SWETZ (N=81) | LLETZ Cone (N=78)
Hysterectomy (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Hysterectomy due to vascular injury
vaginal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Accidental opening of the vaginal mucosa up to near the muscle layer of the bladder.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SWETZ (N=81) | LLETZ Cone (N=78)
Needed general anesthesia (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) — Needed general anesthesia due to some discomfort during the procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No